CLINICAL TRIAL: NCT01676064
Title: Influence of Perioperative Fluid Management on Intraocular Pressure During Hynecologic Laparoscopic Pelvic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0003-12-ZIV
Record Dates: First submitted 2012-08-12; First posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Influence of Perioperative Fluid Regime on Intraocular Pressure During Laparoscopic Gynecologic Surgery
Keywords: intraocular pressure; perioperative fluid; trendelenburg position; laparoscopic gynecologic surgery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- liberal fluid group (Active Comparator): during surgery 7 ml/kg/hr RL during first intraoperative hr, 5 ml/kg/hr for the subsequent hours.After surgery ( PACU) 1,5 ml/kg/hr;After operation ward on the day of surgery 1,5 ml/kg/hr; Postoperative day 1- 1,5 ml/kg/hr RL, oral fluids;Postoperative day 2-oral fluids and solid food according to surgical allowance.
  Interventions: Drug: ringer lactate solution
- restrictive fluid group (Active Comparator): during surgery-RL according to "4-2-1" 4 ml/kg/hr for first 10 kg (=40ml/hr) then 2 ml/kg/hr for next 10 kg (=20ml/hr)then 1 ml/kg/hr for any kg over 20 kg of weight. This always gives 60ml/hr for first 20 kg then you add 1 ml/kg/hr for each kg over 20 kg.
  After surgery (PACU):"4-2-1" rule. After operation ward on the day of surgery 1,5 ml/kg/hr.Postoperative day 1:1,5 ml/kg/hr RL, oral fluids. Postoperative day 2:oral fluids and solid food according to surgical allowance.
  Interventions: Other: restrictive fluid regime

INTERVENTIONS:
Drug: ringer lactate solution
  Arms: liberal fluid group
Other: restrictive fluid regime
  Arms: restrictive fluid group

SUMMARY:
The aim of this study was to quantify the Intraocular Pressure (IOP) changes in patients undergoing laparoscopic hysterectomy at different time points and body positions throughout the procedure, and to explore the influence of perioperative fluid management on the fluctuations of IOP during perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* 50-60 adult female patients,
* ASA physical status I or II,
* scheduled for elective hynecologic laparoscopic pelvic surgery will be included in the study.

Exclusion Criteria:

* patients will be excluded if they are > 70 and < 18 yr of age,
* had have a body weight > 150% of their ideal body weight,
* have acute or chronic eye disease,
* receive any medication known to alter IOP, or
* have any mental illnesses.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
measurements of intraocular pressure during laparoscopic gynecologic surgery a sa function of diffrent perioperative fluid regimes. | 24 hr
IOP will be measured using a Tono-pen® XL by an ophthalmologist who will be unaware of the perioperative fluid administration regimen. | 24 hr

CONTACTS AND LOCATIONS:
Locations (1):
- Sieff Medical Center, Zafed, Israel